CLINICAL TRIAL: NCT01166321
Title: Treatment of Patients With Atypical Meningiomas Simpson Grade 4 and 5 With a Carbon Ion Boost in Combination With Postoperative Photon Radiotherapy: A Phase II Trial
Brief Title: Carbon Ion Radiotherapy for Atypical Meningiomas
Acronym: MARCIE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Prof. Dr. Dr. Jürgen Debus, University Hospital Heidelberg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MARCIE; 2009-016683-36 (EudraCT Number)
Record Dates: First submitted 2010-07-20; First posted 2010-07-21 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Meningioma
Keywords: Atypical Meningioma
MeSH Terms: conditions — Meningioma | interventions — Heavy Ion Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carbon Ion Radiotherapy Boost (Experimental): Carbon Ion Boost to the Macroscopic Tumor visible on contrast-enhanced MR-Imaging
  Interventions: Radiation: Carbon Ion Radiotherapy

INTERVENTIONS:
Radiation: Carbon Ion Radiotherapy — Carbon Ion Boost 18 Gy E in single Fractions of 3 Gy E

SUMMARY:
Treatment standard for patients with atypical or anaplastic meningioma is neurosurgical resection. With this approach, local control ranges between 50 and 70%, depending on resection status. A series or smaller studies has shown that postoperative radiotherapy in this patient population can increase progression-free survival, which translates into increased overall survival. However, meningiomas are known to be radioresistant tumors, and radiation doses of 60 Gy or higher have been shown to be necessary for tumor control.

Carbon ions offer physical and biological characteristics. Due to their inverted dose profile and the high local dose deposition within the Bragg peak precise dose application and sparing of normal tissue is possible. Moreover, in comparison to photons, carbon ions offer an increased relative biological effectiveness (RBE), which can be calculated between 2 and 5 depending on the cell line as well as the endpoint analyzed.

First data obtained within the Phase I/II trial performed at GSI in Darmstadt on carbon ion radiotherapy for patients with high-risk meningiomas has shown safety, and treatment results are promising.

Therefore, in the current Phase II-MARCIE-Study a carbon ion boost will be applied to the macroscopic tumor (gross tumor volume, GTV) in conjunction with photon radiotherapy to the clinical target volume (CTV) in patients with atypical meningiomas after incomplete resection or biopsy.

Primary endpoint is progression-free survival rate, secondary endpoints are overall survival, safety and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed atypical meningioma
* macroscopic tumor after biopsy or subtotal resection
* Simpson Grade 4 or 5
* prior photon radiotherapy to the clinical target volume (CTV) of 48-52 Gy
* beginning of study treatment no later than 12 weeks after surgery
* age ≥ 18 years of age
* Karnofsky Performance Score ≥ 60
* For women with childbearing potential, adequate contraception
* Ability of subject to understand character and individual consequences of the clinical trial
* Written informed consent (must be available before enrolment in the trial)

Exclusion Criteria:

* refusal of the patients to take part in the study
* previous radiotherapy of the brain
* optic nerve sheath meningioma (ONSM)
* time interval of > 12 weeks after primary diagnosis (neurosurgical intervention) and beginning of study treatment
* Patients who have not yet recovered from acute toxicities of prior therapies
* Known carcinoma < 5 years ago (excluding Carcinoma in situ of the cervix, basal cell carcinoma, squamous cell carcinoma of the skin) requiring immediate treatment interfering with study therapy
* Pregnant or lactating women
* Participation in another clinical study or observation period of competing trials, respectively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Progression-free survival at 3 years

SECONDARY OUTCOMES:
Overall Survival | Overall Survival at 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Hopsital Heidelberg, Heidelberg, Germany

REFERENCES:
- [Derived] Combs SE, Edler L, Burkholder I, Rieken S, Habermehl D, Jakel O, Haberer T, Unterberg A, Wick W, Debus J, Haselmann R. Treatment of patients with atypical meningiomas Simpson grade 4 and 5 with a carbon ion boost in combination with postoperative photon radiotherapy: the MARCIE trial. BMC Cancer. 2010 Nov 9;10:615. doi: 10.1186/1471-2407-10-615. PMID 21062428